CLINICAL TRIAL: NCT00225329
Title: Early Labour Support at Home: RCT of Nurse Visits and Telephone Triage
Brief Title: Early Labour Assessment and Support at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C01-0083
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2005-09-23 (Estimated); Status verified 2005-09

CONDITIONS: Latent Phase Labour
Keywords: RCT; intervention study; labour management; assessment
MeSH Terms: interventions — Palliative Care

INTERVENTIONS:
Procedure: Labour assessment and support

SUMMARY:
To determine, among healthy first time mothers who are uncertain as to when to come to hospital in labour, if home visits by obstetrical nurses compared to telephone advice have an impact on reducing cesarean section rate.

DETAILED DESCRIPTION:
Nurses hired by the early labour and support at home (ELASH) study will be situated in the assessment/triage areas of each hospital to recruit subjects for 24 hours per day, seven days per week. After randomization, the study nurse will inform the triage nurses of which arm of the trial the patient has been assigned to. The triage nurses will then provide either of the following interventions.

Telephone Triage In the telephone triage group (standard of care in both hospitals) women will be asked over the phone about the nature and frequency of contractions, presence of bloody show, status of membranes, parity, gestational age, and complications of pregnancy. Based on this information, the nurse will advise the woman as to whether or not to come to hospital. A detailed protocol which outlines telephone documentation, advice-giving and teaching is included in Appendix 1.

Patients who are assessed by telephone not to be in active labour are advised not to come to hospital. In the event that they come anyway, they will receive a hands on assessment (similar to the home visit group) and if assessed not to be in active labour, they will be sent home and encouraged to return home and call in again if they feel that their labour is becoming active.

Home visit by a Nurse Women randomised to the nurse visiting group will be told that a nurse will be leaving the hospital immediately. After obtaining directions to the residence and leaving this information with the charge nurse, the triage nurse will depart. The nursing assessment at home is identical to that which takes place in the triage area of the hospital. It includes a brief history, maternal vital signs, abdominal palpation, auscultation of the fetal heart rate, assessment of contractions, and an examination of the cervix. Comfort measures such as positioning, massage, showering, walking interspersed with resting, use of hot and cold packs, and relaxation techniques will be taught to the woman and her support persons as needed. These will be the same as those outlined in the protocols for telephone triage related to patient teaching. (Appendix 1) Standard advice as outlined in the telephone triage protocol will be given in regard to when to come in to hospital, such as if amniotic fluid is coloured, vaginal bleeding is occurring, contractions were more frequent than 2/10 minutes or lasting longer than 60 seconds or simply too uncomfortable to manage at home. Women in this arm may be visited more than once. The nurse will be in telephone contact with the woman between visits. The nurse will advise the physician of the patient's status from the patient's home. Information related to the home visit is documented on the same form as the telephone documentation with the addition of information from "hands on" assessment, including maternal vital signs, abdominal palpation, fetal heart rate, assessment of cervical dilation and strength of contractions. If remaining at home after the nurse's visit, women will be taught how to contact the nurse on her cellular phone.

ELIGIBILITY:
Inclusion Criteria:

* Pre-registered to deliver at BC Women's or Surrey Memorial Hospital
* Living within a 30-minute drive of the hospital
* Age 16-42
* 37-42 completed weeks of gestation
* Singleton fetus in the vertex position
* Telephone in the home
* Speaks English, Cantonese, Mandarin or Punjabi
* Nulliparous

Exclusion Criteria:

* Women whose primary caregivers are midwives. (women who are receiving midwifery care are excluded because midwives routinely visit their clients in early labour at home. At present there are only 30 midwife-attended births per month in both hospitals combined.)
* Women whose prenatal record (forwarded to the hospital at 36 weeks) documents abnormalities of the placenta, diabetes, either gestational or pre-existing, maternal cardio-vascular or renal dysfunction, fetal anomalies or abnormal amniotic fluid volumes, or any other concern documented on the prenatal form which would preclude the parturient labouring in the latent phase of labour at home.

Ages: 16 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1466
Dates: Start 2001-09; Study Completion 2004-08

PRIMARY OUTCOMES:
Rate of cesarean section

SECONDARY OUTCOMES:
• rates of admission to the delivery suite of women in the latent phase of labour (< 3 cm of cervical dilatation)
• augmentation of labour, either surgically or medically
• use of narcotic given intravenously or intramuscularly in labour
• use of epidural analgesia.
• Newborn Apgar scores at 1 and 5 minutes
• need for Intermittent Positive Pressure Ventilation by mask or endotracheal tube at birth
• newborn admission to level II or III nursery

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Janssen, PhD, Principal Investigator — University of British Columbia